CLINICAL TRIAL: NCT03326596
Title: Prevention of Postpartum Hemorrhage With Tranexamic Acid (TXA)
Brief Title: Prevention of Postpartum Hemorrhage With TXA
Acronym: TXA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI retired from Navy 2018
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sidrah Malik, Program Director, Obstetrics & Gynecology Residency, United States Naval Medical Center, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMCSD.2017.0034
Record Dates: First submitted 2017-10-10; First posted 2017-10-31 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Postpartum Hemorrhage
Keywords: Hemorrhage; Tranexamic acid (TXA); Estimated Blood Loss (EBL)
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ProphylacticTranexamic Acid (Experimental): Once consented, patients to receive 1000mg/10ml normal saline infusion of TXA with the delivery of the infant's anterior shoulder.
  Interventions: Drug: Tranexamic Acid 1000 mg/10ml normal saline infusion

INTERVENTIONS:
Drug: Tranexamic Acid 1000 mg/10ml normal saline infusion — Infusion of Tranexamic Acid (Cyklokapron) to all consented women with the delivery of the anterior shoulder of the infant
  Other Names: Cyklokapron

SUMMARY:
Hemorrhage remains the leading cause of maternal death worldwide. Tranexamic acid has been shown to reduce rates of hemorrhage when given prophylactically prior to cesarean delivery. It has also been shown to be an effective treatment in response to hemorrhage after a vaginal delivery. The aim of this study is to assess the impact of TXA on hemorrhage rates when given prophylactically prior to all deliveries.

DETAILED DESCRIPTION:
Hemorrhage remains the leading cause of maternal mortality worldwide. In a 2014 systematic analysis of the causes of maternal death, the World Health Organization (WHO) noted that even in the face of interventions developed to actively manage the third stage of labor, 27.1% of maternal deaths were directly attributable to excessive blood loss.

Risk factors for postpartum hemorrhage (PPH) have been identified, but the majority of cases occur in low risk women. As such, the routine use of oxytocin in the third stage of labor is recommended in all women and has been well documented to reduce the risk of excessive blood loss. Uterotonics such as methylergonovine, 15-methyl PGF2α and misoprostol have shown to be particularly useful adjuncts as decreased uterine tone is the most common etiology of blood loss. More recently, tranexamic acid (TXA) has been shown to be efficacious in the prevention of postpartum hemorrhage in certain cohorts.

Tranexamic acid exerts its effect through the binding of plasmin and subsequent inhibition of fibrin degradation. It is regarded as pregnancy category B by the Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female presenting to Navy Medical Center San Diego for delivery
* Able to speak and understand English
* Planning to deliver at NMCSD

Exclusion Criteria:

* Age less than 18 years
* Unable to speak or understand English
* Not planning to deliver at NMCSD
* Planned cesarean hysterectomy
* Current anticoagulant use
* Current subarachnoid hemorrhage
* Any active/current intravascular clotting (i.e. venous thromboembolic events)
* Patients with a hypersensitivity to TXA or any of the ingredients
* Personal history of venous or arterial thrombotic events
* Conditions that predispose patients to thromboembolic events (e.g. thrombophilias, autoimmune diseases such as lupus, active cancer, congestive heart failure, family history of thrombosis in a first degree relative at age < 30 years) due to increased risk of thrombosis
* Patients taking factor IX complex concentrates or anti-inhibitor coagulant concentrates (e.g. FEIBA NF)
* Eclampsia or seizure disorder because the use of tranexamic acid has been associated with postoperative seizures
* Patients with a baseline creatinine 1.2 or higher, history of renal insufficiency, or renal disease because of the risk of toxicity in patients with preexisting disease
* Patients with frank hematuria because ureteral obstruction due to clot formation has been reported in patients with upper urinary tract bleeding who were treated with tranexamic acid
* Patients with active or history of retinal diseases as cases of central retinal artery and central retinal vein obstruction have been reported in patients treated with intravenous tranexamic acid
* Patients with acquired defective color vision

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of postpartum hemorrhage | Up to six weeks from date of delivery
  Postpartum hemorrhage

SECONDARY OUTCOMES:
Postpartum blood loss | Up to six weeks from date of delivery
  Estimated blood loss (EBL)
Percent decrease in hematocrit | 6 hours after hemorrhage event and as clinically indicated up to six weeks from date of delivery
  Hematocrit percentage
Number of units of packed red blood cells transfused | Up to six weeks from date of delivery
  Number of units of packed red blood cells transfused
Number of units of platelets transfused | Up to six weeks from date of delivery
  Number of units of platelets transfused
Number of units of fresh frozen plasma transfused | Up to six weeks from date of delivery
  Number of units of fresh frozen plasma transfused
Number of units of cryoprecipitate transfused | Up to six weeks from date of delivery
  Number of units of cryoprecipitate transfused
Amount of methylergonovine administered | Up to six weeks from date of delivery
  Amount of methylergonovine administered
Amount of 15-methyl prostaglandin F2(PGF2) administered | Up to six weeks from date of delivery
  Amount of 15-methyl prostaglandin F2(PGF2) administered
Amount of misoprostol administered | Up to six weeks from date of delivery
  Amount of misoprostol administered
Amount of oxytocin administered | Up to six weeks from date of delivery
  Amount of oxytocin administered
Exploratory laparotomy following vaginal delivery due to hemorrhage | Up to six weeks from date of delivery
  Exploratory laparotomy, no hysterectomy
Exploratory laparotomy following cesarean delivery due to hemorrhage | Up to six weeks from date of delivery
  Exploratory laparotomy, no hysterectomy
Hysterectomy | Up to six weeks from date of delivery
  Number of hysterectomies performed as a result of postpartum hemorrhage
Intensive Care Unit (ICU) admission | Up to six weeks from date of delivery
  Number of subjects admitted to Intensive Care Unit diagnosed with postpartum hemorrhage
Maternal thromboembolic events | up to six weeks from date of delivery
  Incidence of maternal thromboembolic events
Diagnosis of intraventricular hemorrhage in the neonate | Up to six weeks from date of delivery
  Neonatal outcome intraventricular hemorrhage
Diagnosis of anemia in the neonate | Up to six weeks from date of delivery
  Neonatal outcome anemia
Diagnosis of disseminated intravascular coagulation (DIC) in the neonate | Up to six weeks from date of delivery
  Neonatal outcome DIC
Diagnosis of neonatal sepsis | Up to six weeks from date of delivery
  Neonatal outcome sepsis
Diagnosis of hypoxic-ischemic encephalopathy (HIE) in the neonate | Up to six weeks from date of delivery
  Neonatal outcome HIE
Diagnosis of a seizure disorder in the neonate | Up to six weeks from date of delivery
  Neonatal outcome seizure disorder
Diagnosis of arrhythmia in the neonate | Up to six weeks from date of delivery
  Neonatal outcome arrhythmia
Diagnosis of heart failure in the neonate | Up to six weeks from date of delivery
  Neonatal outcome heart failure
Diagnosis of renal failure in the neonate | Up to six weeks from date of delivery
  Neonatal outcome renal failure
Diagnosis of hepatic failure in the neonate | Up to six weeks from date of delivery
  Neonatal outcome hepatic failure
Diagnosis of thromboembolic events in the neonate | Up to six weeks from date of delivery
  Neonatal outcome thromboembolic event
Maternal mortality | Up to six weeks from date of delivery
  Incidence of maternal mortality
Additional tranexamic acid administered | Up to six weeks from date of delivery
  Additional tranexamic acid administered
Rate of Bakri/balloon tamponade use | Up to six weeks from date of delivery
  Bakri/balloon tamponade use

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Farrell, MD, Principal Investigator — United States Naval Medical Center, San Diego,CA
Locations (1):
- Navy Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Zelop CM. Postpartum hemorrhage: becoming more evidence-based. Obstet Gynecol. 2011 Jan;117(1):3-5. doi: 10.1097/AOG.0b013e318202ec9a. No abstract available. PMID 21173639
- [Background] WHO Recommendations for the Prevention and Treatment of Postpartum Haemorrhage. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK131942/ PMID 23586122
- [Result] Sentilhes L, Lasocki S, Ducloy-Bouthors AS, Deruelle P, Dreyfus M, Perrotin F, Goffinet F, Deneux-Tharaux C. Tranexamic acid for the prevention and treatment of postpartum haemorrhage. Br J Anaesth. 2015 Apr;114(4):576-87. doi: 10.1093/bja/aeu448. Epub 2015 Jan 8. PMID 25571934
- [Result] Novikova N, Hofmeyr GJ, Cluver C. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2015 Jun 16;2015(6):CD007872. doi: 10.1002/14651858.CD007872.pub3. PMID 26079202
- [Result] Wang HY, Hong SK, Duan Y, Yin HM. Tranexamic acid and blood loss during and after cesarean section: a meta-analysis. J Perinatol. 2015 Oct;35(10):818-25. doi: 10.1038/jp.2015.93. Epub 2015 Jul 30. PMID 26226243
- [Result] Simonazzi G, Bisulli M, Saccone G, Moro E, Marshall A, Berghella V. Tranexamic acid for preventing postpartum blood loss after cesarean delivery: a systematic review and meta-analysis of randomized controlled trials. Acta Obstet Gynecol Scand. 2016 Jan;95(1):28-37. doi: 10.1111/aogs.12798. Epub 2015 Nov 12. PMID 26698831
- [Result] Ker K, Shakur H, Roberts I. Does tranexamic acid prevent postpartum haemorrhage? A systematic review of randomised controlled trials. BJOG. 2016 Oct;123(11):1745-52. doi: 10.1111/1471-0528.14267. Epub 2016 Aug 24. PMID 27558956
- [Result] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Result] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Result] Bouet PE, Ruiz V, Legendre G, Gillard P, Descamps P, Sentilhes L. Policy of high-dose tranexamic acid for treating postpartum hemorrhage after vaginal delivery. J Matern Fetal Neonatal Med. 2016;29(10):1617-22. doi: 10.3109/14767058.2015.1056731. Epub 2015 Jun 29. PMID 26118386
- [Result] Sujata N, Tobin R, Kaur R, Aneja A, Khanna M, Hanjoora VM. Randomized controlled trial of tranexamic acid among parturients at increased risk for postpartum hemorrhage undergoing cesarean delivery. Int J Gynaecol Obstet. 2016 Jun;133(3):312-5. doi: 10.1016/j.ijgo.2015.09.032. Epub 2016 Feb 16. PMID 26952346

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03326596/Prot_SAP_001.pdf
  • Study Protocol: Protocol Cover Page (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03326596/Prot_002.pdf
  • Informed Consent Form: Informed Consent (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03326596/ICF_000.pdf
  • Informed Consent Form: Informed Consent Cover Page (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03326596/ICF_003.pdf